CLINICAL TRIAL: NCT02196766
Title: BIOCLEAN FIRST CARE EX in Combination With Biofinity Lens: A Two Week Crossover Study
Brief Title: BIOCLEAN FIRST CARE EX in Combination With Biofinity Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CVJ-EX-MKTG-1818
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — comfilcon A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioclean First Care EX combo, then Aosept Clearcare combo (Active Comparator): Subjects dispensed Bioclean First Care EX / comfilcon A combination then crossed over to the Aosept Clearcare / comfilcon A combination.
  Interventions: Other: Bioclean First Care EX / comfilcon A; Other: Aosept Clearcare / comfilcon A
- Aosept Clearcare combo, then Bioclean First Care EX combo (Active Comparator): Subjects dispensed Aosept Clearcare / comfilcon A combination then crossed over to the Bioclean First Care EX / comfilcon A combination.
  Interventions: Other: Bioclean First Care EX / comfilcon A; Other: Aosept Clearcare / comfilcon A

INTERVENTIONS:
Other: Bioclean First Care EX / comfilcon A — Subjects dispensed Bioclean First Care EX / comfilcon A combination then crossed over to the alternate combination.
Other: Aosept Clearcare / comfilcon A — Subjects dispensed Aosept Clearcare / comfilcon A combination then crossed over to the alternate combination.

SUMMARY:
To determine if patients are unreactive to the lens care solution / Biofinity combination.

DETAILED DESCRIPTION:
To determine if patients are unreactive to the lens care solution / Biofinity combination in this cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Is over 18 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is currently an adapted spherical soft CL wearer
* Has a CL spherical prescription between - 0.25 and - 12.00 (inclusive)
* Has less than 1.00D spectacle cylinder in each eye.
* Is correctable to a visual acuity of 20/20 or better in both eyes
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Is willing to comply with the wear schedule (at least 40 hrs per week)
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has never worn contact lenses before.
* Currently wears rigid gas permeable contact lenses.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has a CL prescription outside the range of - 0.25 to -12.00D
* Has a spectacle cylinder greater than -0.75D of cylinder in either eye.
* Has best corrected spectacle distance vision worse than 20/20 in either eye.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion
* Has persistent, clinically significant corneal or conjunctival staining
* Has active neovascularization or any central corneal scars.
* Is aphakic.
* Is pregnant or lactating.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taku Muraoka, OD, Study Director — Director Professional Services, CVI Japan
Locations (3):
- Japan (3):
  - Kokama Eye Clinic, Joyo-shi, Kyoto
  - Higashihara Clinic, Kameoka, Kyoto
  - Dougenzaka Ioti Eye Clinic, Shibuya-ku, Tokyo-to

RESULTS

PARTICIPANT FLOW:
Groups:
- Bioclean First Care EX Combo, Then Aosept Clearcare Combo; Aosept Clearcare Combo First,Then Bioclean First Care EX Combo: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
Period: First Intervention (7 Days)
Arm/Group | Bioclean First Care EX Combo, Then Aosept Clearcare Combo | Aosept Clearcare Combo First,Then Bioclean First Care EX Combo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Bioclean First Care EX Combo, Then Aosept Clearcare Combo | Aosept Clearcare Combo First,Then Bioclean First Care EX Combo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall participants group prior to randomization of study lens pairs and solution.
Groups:
- Bioclean First Care EX / Aosept Clearcare / Comfil: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
Arm/Group | Bioclean First Care EX / Aosept Clearcare / Comfil
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Region of Enrollment [Number; unit: participants]
  Japan | 30

OUTCOME MEASURES:

1. Primary Outcome: Ocular Health - Corneal Staining
Description: Corneal staining for each combination was assessed by slit lamp at 1 week. (Grade 0-4; 0=normal, 1=trace, 2=mild, 3=moderate, 4= severe).
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Bioclean First Care EX / Comfilcon A: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
  Bioclean First Care EX / comfilcon A: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
- Aosept Clearcare / Comfilcon A: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
  Aosept Clearcare / comfilcon A: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Normal | 38 | 35
  Trace | 18 | 20
  Mild | 4 | 5
  Moderate | 0 | 0
  Severe | 0 | 0

2. Secondary Outcome: Stinging Sensation Right After Insertion (Subjective Rating)
Description: Subjective rating of stinging sensation for the combinations is assessed at baseline. (Scale 0-10; 0=difficult to wear, 10=no sensation at all).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale | 9.5 (1.1) | 9.4 (1.2)

3. Secondary Outcome: Burning Sensation Right After Insertion (Subjective Rating)
Description: Subjective rating of burning sensation right after insertion for each combination assessed at baseline. (Scale 0-10; 0=difficult to wear, 10=no sensation at all).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Number analyzed (Participants) | 30 | 30
units on a scale | 9.5 (1.1) | 9.4 (1.2)

4. Primary Outcome: Ocular Health - Conjunctival Redness
Description: Conjunctival redness for each combination was assessed by slit lamp at 1 week. (Grade 0-4; 0=normal, 1=trace, 2=mild, 3=moderate, 4= severe).
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Normal | 40 | 40
  Trace | 20 | 20
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0

5. Primary Outcome: Ocular Health - Limbal Redness
Description: Limbal redness for each combination was assessed by slit lamp at 1 week. (Grade 0-4; 0=normal, 1=trace, 2=mild, 3=moderate, 4= severe).
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Normal | 49 | 47
  Trace | 11 | 12
  Mild | 0 | 1
  Moderate | 0 | 0
  Severe | 0 | 0

6. Primary Outcome: Ocular Health - Papillary Conjunctivitis
Description: Papillary conjunctivitis for each combination was assessed by slit lamp at 1 week. (Grade 0-4; 0=normal, 1=trace, 2=mild, 3=moderate, 4= severe).
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Normal | 52 | 51
  Trace | 7 | 8
  Mild | 1 | 1
  Moderate | 0 | 0
  Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: From dispense up to two weeks for study lenses with both study lens care solutions
Groups:
- Aosept Clearcare / Comfilcon A: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
  Bioclean First Care EX / comfilcon A: Subjects dispensed either Bioclean First Care EX / comfilcon A combination or Aosept Clearcare / comfilcon A combination and then crossover to the alternate combination.
Arm/Group | Bioclean First Care EX / Comfilcon A | Aosept Clearcare / Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.